CLINICAL TRIAL: NCT05812547
Title: A Novel Device for Gestational Diabetes Control, a Randomized Control Trial
Brief Title: A Novel Device for Gestational Diabetes Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0572-21-RMB CTIL
Record Dates: First submitted 2022-11-22; First posted 2023-04-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: This will be an open label parallel group 1:1 randomized-controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Lumen group (Experimental): subjects will use the Lumen device and mobile phone application, which will guide them once a day after the night fast regarding their daily diet, sleep, and routines according to their Lumen measurements. Subjects will need Google Fit (Android) or Apple Health Kit (iOS) and will be encouraged to communicate with a study investigator via the app during the entirety of the study to resolve technical questions about the device and data collection
  Interventions: Device: Lumen
- The control group (Active Comparator): The control group will use a mobile app to keep track of their glucose levels and will be managed in accordance with the common guidelines for GDM management. Participants of both groups will measure their fasting blood glucose levels and their postprandial blood glucose levels and record it in their mobile app
  Interventions: Other: Glucose monitoring mobile app

INTERVENTIONS:
Device: Lumen — subjects will use the Lumen device and mobile phone application, which will guide them once a day after the night fast regarding their daily diet, sleep, and routines according to their Lumen measurements. Subjects will need Google Fit (Android) or Apple Health Kit (iOS) and will be encouraged to communicate with a study investigator via the app during the entirety of the study to resolve technical questions about the device and data collection.
  Arms: The Lumen group
Other: Glucose monitoring mobile app — The control group will use a designated glucose monitoring mobile app to record their glucose levels
  Arms: The control group

SUMMARY:
Rationale of the study: Gestational diabetes mellitus (GDM) is very common and the rate of women suffering from it expected to increase in the next years. It is associated with maternal and fetal morbidity and the risk is correlated to the patient's degree of glucose control which can be achieved through a change in lifestyle or medication. Several studies have demonstrated the effectiveness of mobile apps in improving obstetric outcomes in GDM. In addition, the LUMEN device is a breathing device that produces dietary and exercise recommendations based on CO2 levels and improves metabolic parameters in patients with type 2 diabetes. No work has been done on its effectiveness in treating GDM. Aims of the study: Comparison of metabolic outcomes in women with gestational diabetes, with or without the use of LUMEN app. Design: This will be an open label parallel group 1:1 randomized-controlled trial Methods: the investigators will recruit women diagnosed with GDM. The women will be randomized to the intervention arm that will use the LUMEN device and app or to the control arm that will use a free mobile tracking app. The women will be required to monitor their blood sugar levels daily and to have GDM follow-up in the feto-maternal outpatient clinic, as is customary in GDM. After the birth, the maternal and neonatal outcome will be recorded. Based on past research data, a recruitment of 170 is needed to demonstrate a 16.7% decrease in insulin use to balance diabetes, with α = 0.05 and β = 80.

DETAILED DESCRIPTION:
Objective The aim of the study is to examine the effect of using Lumen on metabolic parameters and anthropometric variables in patients with gestational diabetes mellitus. Aims and hypotheses Primary aim: To evaluate the rate of progression from GDM-A1 to GDM-A2 between the groups.

Secondary aim: To evaluate the efficacy of Lumen on metabolic parameters, obstetric outcomes, and neonatal outcomes. Hypothesis: the investigators expect that using Lumen would reduce the rate of progression from GDM-A1 to GDM- A2. Methods Design This will be an open label parallel group 1:1 randomized-controlled trial. Participants The study will include up to 170 women diagnosed with GDM. GDM will be defined according to current ACOG (The American College of Obstetricians and Gynecologists) guidelines. A positive glucose challenge test at 24-28 weeks' gestation followed by at least two pathological values in oral glucose challenge or one pathological value and at least one additional risk factor for GDM (a first family member diagnosed with type 2 DM, obesity, history of GDM).

Women in both groups it will use a glucometer and will be instructed in the use of the device. Use will include puncture of the fingertip to obtain a drop of blood and use of a suitable probe to obtain a sugar measurement.

Eligibility criteria

Inclusion criteria:

1. Gravidas aged 18-45 years
2. Singleton pregnancy
3. Diagnosed with GDM in current pregnancy
4. First visit to high-risk pregnancy clinic is no late than 32 weeks' gestation
5. Not treated with diabetes-related medications

Exclusion criteria:

Medications:

1. Insulin and medications for glycemic control
2. Antipsychotics
3. Diuretics
4. Corticosteroids
5. Oncologic treatment

Version 4.0 , 24/05/2022 0572-21-RMB

5

Conditions:

1. Previous diagnosis of diabetes
2. Renal disease
3. Hepatic disease

Personal requirements:

1. Inability to read and understand English
2. Inability to use a smartphone
3. Any issues arise with using the Lumen device and application
4. Aerobic exercise > 3 times per week Recruitment Women with GDM will be recruited via clinical referrals from the feto-maternal outpatient clinic or the feto-maternal unit in Rambam medical center (RMC) Intervention All the participants will be under regular follow-up of the treating obstetrician in the feto-maternal outpatient clinic. After the diagnosis of GDM the patients (of both groups) will be instructed regarding recommended diet and glucose monitoring as accustomed in our department. After randomization to the lumen group, subjects will use the Lumen device and mobile phone application, which will guide them once a day after the night fast regarding their daily diet, sleep, and routines according to their Lumen measurements. Subjects will need Google Fit (Android) or Apple Health Kit (iOS) and will be encouraged to communicate with a study investigator via the app during the entirety of the study to resolve technical questions about the device and data collection. The control group will use the glucose buddy app and will be managed in accordance with the common guidelines for GDM management. Participants of both group will measure their fating blood glucose levels and their postprandial blood glucose levels and record it in their mobile app.

ELIGIBILITY:
Inclusion Criteria:

1. Gravidas aged 18-45 years
2. Singleton pregnancy
3. Diagnosed with GDM in current pregnancy
4. First visit to high-risk pregnancy clinic is no late than 32 weeks' gestation
5. Not treated with diabetes-related medications

Exclusion Criteria:

-

Medications:

1. Insulin and medications for glycemic control
2. Antipsychotics
3. Diuretics
4. Corticosteroids
5. Oncologic treatment

Conditions:

1. Previous diagnosis of diabetes
2. Renal disease
3. Hepatic disease

Personal requirements:

1. Inability to read and understand English
2. Inability to use a smartphone
3. Any issues arise with using the Lumen device and application
4. Aerobic exercise > 3 times per week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the average change in blood glucose levels with the use the Lumen device | From date of randomization until the date delivery, assessed up to 4 months
  The blood glucose levels will be recorded and the average levels will be compared between the groups

SECONDARY OUTCOMES:
to compare the maternal age | From date of randomization until the date delivery, assessed up to 4 months
  maternal age in years
to compare the gestational age at delivery | From date of randomization until the date delivery, assessed up to 4 months
  gestational age at delivery in weeks
to compare the parity between the groups | From date of randomization until the date delivery, assessed up to 4 months
  parity
to compare the rate of family history of DM | From date of randomization until the date delivery, assessed up to 4 months
  family history of DM
to compare the rate of chronic hypertension | From date of randomization until the date delivery, assessed up to 4 months
  reported chronic hypertension
to compare smoking status | From date of randomization until the date delivery, assessed up to 4 months
  smoking status in medical records
to compare baseline fertility characteristics | From date of randomization until the date delivery, assessed up to 4 months
  Need for assisted reproductive technology
to compare baseline metabolic parameters | From date of randomization until the date delivery, assessed up to 4 months
  fasting glucose obtained at first trimester, values of glucose challenge test (GCT) and oral glucose tolerance test (OGTT), hemoglobin A1C (HbA1C) upon diagnosis
to compare baseline educational status | From date of randomization until the date delivery, assessed up to 4 months
  years of education
to compare the level of physical activity | at the date of randomization
  level of physical activity as reported by the patients
to compare baseline body mass index between the groups | at the date of randomization
  patient's body mass index (BMI)
To compare the Gestational age at delivery | at the date if delivery
  Gestational age at delivery in weeks
to compare the mode of onset of labor | at the date if delivery
  mode of onset of labor (medical or surgical)
to compare the rate of of preeclampsia or gestational hypertension | From date of randomization until the date delivery, assessed up to 4 months
  the presence of preeclampsia or gestational hypertension
to compare the rate of polyhydramnios | From date of randomization until the date delivery, assessed up to 4 months
  polyhydramnios (amniotic fluid index > 95th percentile for gestational age)
To compare the rate of antenatal corticosteroids administration | From date of randomization until the date delivery, assessed up to 4 months
  Antenatal corticosteroids administration
To evaluate the efficacy of Lumen on mode of delivery | At the date of delivery
  mode of delivery
To evaluate the efficacy of Lumen on shoulder dystocia rate | At the date of delivery
  shoulder dystocia as reported in medical records
To compare the rate of episiotomy | At the date of delivery
  the use of episiotomy
To evaluate the change it the rate of obstetric anal sphincter injuries | At the date of delivery
  Rate of obstetric anal sphincter injuries
To evaluate the change in birthweight | At the date of delivery
  Birth weight in grams
To evaluate the change in neonatal death rate | from the date of delivery and up to 1 month from delivery
  neonatal death rate
To evaluate the change in neonatal length of stay | from the date of delivery and up to 1 month from delivery
  neonatal length of stay in days
To evaluate the change in hypoglycemia of the newborn | from the date of delivery and up to 1 month from delivery
  hypoglycemia of the newborn is defined as blood glucose levels below 40
To evaluate the change in respiratory morbidity | from the date of delivery and up to 1 month from delivery
  respiratory morbidity
To evaluate the change in need for phototherapy | from the date of delivery and up to 1 month from delivery
  Need for phototherapy
To evaluate the change in need for neonatal intensive care unit (NICU) admission | from the date of delivery and up to 1 month from delivery
  neonatal intensive care unit (NICU) admission

IPD SHARING:
Plan to Share IPD: Undecided